CLINICAL TRIAL: NCT05436119
Title: Select Nutrient and Gene Variant Analysis in a Targeted Diet and Lifestyle Intervention Reduces Preterm Birth (SNGLI-PTB)
Brief Title: Select Nutrient and Gene Variant Analysis in a Targeted Diet and Lifestyle Intervention Reduces Preterm Birth
Acronym: SNGLI-PTB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: GrowBaby Life Project (Other)
Collaborators: Metagenics, Inc. (Industry); OmegaQuant, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GrowBaby/Molina PIP 2022
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Premature Birth; Pre-Eclampsia; Small for Gestational Age Infant
Keywords: Nutrition; Lifestyle; Probiotics; Gene variants; Medicaid
MeSH Terms: conditions — Premature Birth; Pre-Eclampsia | interventions — Diet; Probiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dried blood spot analyzed for 44 relevant gene variants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GrowBaby: All pregnant women presenting at < 19 weeks EGA for prenatal care covered by Molina Health of Nevada MCO will be offered the GrowBaby group nutrition and lifestyle program. Primary and secondary outcomes of those who opt out of the program will be compared to those who opt in. Additionally, all women who develop primary or secondary outcomes in the GrowBaby arm will be compared to those who do not develop primary or secondary outcomes (nested case-control). Outcomes will be compared locally, regionally and nationally within the Medicaid population, as well.
  Interventions: Dietary Supplement: GrowBaby

INTERVENTIONS:
Dietary Supplement: GrowBaby — Virtual group educational visits will cluster women in the same trimester of pregnancy teaching trimester-specific diet and lifestyle modification, further customized to the individual using limited micronutrient and gene variant analysis. Each woman will receive base multi-nutrient and probiotic supplementation with customization if identified needs cannot be met with diet and lifestyle modification alone.
  Other Names: Dietary; Probiotic; Behavioral

SUMMARY:
Preterm birth (PTB) rates in the US are among the highest in wealthy nations across the globe, and they are particularly high in our most socio-economically disadvantaged populations. PTB increases lifelong morbidity and mortality at significant economic cost. In addition to neonates born too early, small for gestational infants predict the greatest risk for chronic disease in the neonate (F1 generation) through adulthood. Single lifestyle, nutrient, or medical interventions intended to reduce PTB have produced mixed results, but combined micronutrient interventions appear more successful. The investigators experienced a reduced preterm birth rate and combined preeclampsia, gestational diabetes and small for gestational age rate in a 50% Medicaid population by providing targeted micro/macronutrient, genomic and lifestyle evaluation with personalized intervention in a trimester-by-trimester group educational setting (1). The model requires validation in more diverse populations.

This study will be applied in a 100% Medicaid population with greater ethnic diversity. Participation will be voluntary, offered to all pregnant participants enrolling at 18 weeks gestation or earlier with the comparator group being those participants who decline the intervention. The study population will receive targeted biomarker evaluation including serum 25-OH D, zinc and carnitine levels, dried blood spot omega 3 fatty acids and select gene variant analysis. Virtual group nutrition and lifestyle education visits conducted by the nutritionist cluster participants in the same trimester allowing for personalization of the nutrition and lifestyle plan based on the data collected and adapted to the specific needs of the trimester. Each study participant will receive individualized nutrient supplementation and probiotic supplementation. Anticipated performance improvement endpoints are significant reduction of preterm birth and combined incidence of preeclampsia, gestational diabetes, small for gestational age, neonatal morbidities and related health care expenses. The investigators will explore gene variants' role in directing nutrition, lifestyle and toxic exposure interventions and in predicting adverse maternal and neonatal outcomes.

DETAILED DESCRIPTION:
Hypothesis:

• Diet and lifestyle education with diet and lifestyle modification will significantly decrease the incidence of preterm birth (PTB).

Secondary Hypothesis:

• Diet and lifestyle education and modification refined by limited genomics and nutrient biomarkers will significantly decrease the incidence of preeclampsia (preE), gestational diabetes mellitus (GDM), small for gestational age (SGA) and large for gestational age (LGA) neonates, and neonatal hospitalizations within the first 2 weeks of life.

Exploratory Hypotheses:

* A gene variant pattern will emerge that predicts PTB.
* A gene variant pattern will emerge that predicts preE, GDM, SGA, and LGA.

Goals:

* Ascertain PTB rates for both intervention and non-intervention groups.
* Ascertain preE, GDM, SGA, LGA, and neonatal hospitalization rates for both groups.
* Correlate diet and lifestyle education and modification refined by limited genomics and micronutrient biomarkers with reduced primary and secondary outcomes.
* Reduce related net healthcare costs.

Methods:

• Prospective longitudinal observational cohort with nested case-control study.

Relevance:

* Determine whether diet and lifestyle education and modification refined by trimester and by limited genomics and micronutrient biomarkers applied to a 100% Medicaid population is associated with reduced rates of PTB, preE, GDM, SGA, LGA, and neonatal hospitalizations.
* Determine whether the reduction in pregnancy and neonatal morbidities is associated with a reduction in related net health care costs.
* Explore predictive capability of limited genomics panel in a 100% Medicaid population.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* gestational age < 19 weeks at time of enrollment
* Health care coverage through Molina Health of Nevada MCO
* Residing in the state of Nevada
* Signed consent

Exclusion Criteria:

* Not pregnant
* Gestational age > 19 weeks at time of enrollment
* Health care coverage not through Molina
* Living outside the state of Nevada
* No signed consent or unable to give informed consent

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The study population is derived from pregnant women managed at OB/GYN Clinics in Southern Nevada whose health care is covered by Molina Health Nevada MCO.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Preterm Birth < 37 weeks EGA | At conclusion of pregnancy
  Evaluating the percentage of preterm birth in each group, further divided by delivery < 28 weeks, 28 to <= 32 weeks, 32 to <= 36 weeks, and 36 to <= 37 weeks.

SECONDARY OUTCOMES:
Preeclampsia | At conclusion of pregnancy
  Evaluating the percentage of preeclampsia, condition defined by ACOG standards
Gestational diabetes mellitus(GDM) | At conclusion of pregnancy
  Evaluating the percentage of GDM in each group, condition defined by ACOG standards
Small for gestational age infant (SGA) | At conclusion of pregnancy
  Evaluating the percentage of SGA in each group, condition defined by APP standards.
Large for gestational age infant (LGA) | At conclusion of pregnancy
  Evaluating the percentage of LGA in each group, condition defined by APP standards.
Neonatal hospitalization within 2 weeks of delivery | 8 weeks postpartum
  Evaluating the percentage of neonatal hospitalization within 2 weeks of delivery in each group

OTHER OUTCOMES:
Gene variant pattern analysis | At 20 weeks EGA
  Evaluating association of gene variant patterns with primary and secondary outcomes in each group, and in the nested case control subset

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stone, MD, Study Chair; Leslie P Stone, MD, Principal Investigator
Locations (1):
- Women's Health Associates of Nevada (WHAsN), Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. At completion of the study all the data will be de-identified and grouped for purposes of analysis and publication.

REFERENCES:
- [Background] Stone LP, Stone PM, Rydbom EA, Stone LA, Stone TE, Wilkens LE, Reynolds K. Customized nutritional enhancement for pregnant women appears to lower incidence of certain common maternal and neonatal complications: an observational study. Glob Adv Health Med. 2014 Nov;3(6):50-5. doi: 10.7453/gahmj.2014.053. PMID 25568832